CLINICAL TRIAL: NCT06651710
Title: Effects of Zynamite® on Cognitive Function and Mood in University Students
Brief Title: Zynamite® in Cognition and Mood in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: University
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: University Student

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (No Intervention)
- Zynamite® soluble 100mg (Experimental)
  Interventions: Other: Zynamite
- Zynamite® soluble 150mg (Experimental)
  Interventions: Other: Zynamite

INTERVENTIONS:
Other: Zynamite — Two doses of Mangifera indica leaf extract in its soluble form, Zynamite® S, 100 mg of which 60 mg is mangiferin and 150 mg of which 90 mg is mangiferin, will be tested against a placebo. On the day of the test, the supplements will be administered 30 minutes before the start of the test. The supplements or placebo will be administered in cellulose capsules or similar and accompanied by a glass of water.
  Arms: Zynamite® soluble 100mg; Zynamite® soluble 150mg

SUMMARY:
This study examines the effects of a single dose of ZynS on cognitive function (memory, concentration, attention, and mental agility) in college students and will test the efficacy of this treatment on mood (anger, fatigue, vigor, agreeableness, tension, and depression).

ELIGIBILITY:
Inclusion Criteria:

* Be an active undergraduate or graduate student
* Be between 18 and 25 years of age
* Be healthy and free of any relevant medical condition or disease.

Exclusion Criteria:

* Suffer from chronic diseases such as asthma, type 1 diabetes, thyroid diseases (such as hypothyroidism or hyperthyroidism), autoimmune disorders (such as Crohn's disease) and psychiatric conditions such as anxiety disorders, major depression, eating disorders (anorexia, bulimia), attention deficit hyperactivity disorder (ADHD), among others; ii) Pregnancy or breastfeeding.
* Known intolerance, hypersensitivity or allergies to any of the ingredients of the products under investigation;
* Intestinal absorption problems, as well as learning difficulties, dyslexia, eye problems or color blindness;
* Intake of psychoactive substances or medications that may influence the results of the study, such as consuming >500 mg of caffeine per day (>6 cups of 150 ml filtered coffee) and/or alcohol;
* Having comprehension or communication difficulties that prevent full understanding of the informed consent or effective participation in the study, such as autism spectrum disorders, aphasia, or intellectual disability.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
del POMS (Profile Of Mood States) | Up to fourteen days
  It has a total of 6 subscales: tension (score range, 0-36), depression (score range, 0-60), anger (score range, 0-48), fatigue (score range, 0-28), vigor (score range, 0-32), and confusion (score range, 0-28), and a total mood disturbance (score range, -32 to 200). Each of the questions will be scored from 0 (not at all) to 4 (very much so). The total mood disturbance score is calculated by summing the five negative subscale scores (tension, depression, anger, fatigue, and confusion) and subtracting the vigor score. Higher scores for the total mood disturbance score indicate a greater degree of mood disturbance.
Rey Auditory Verbal Learning Test (RAVLT) | Up to fourteen days
  The Rey Auditory Verbal Learning Test (RAVLT) is a neuropsychological test used to assess short- and long-term memory. The structure of the RAVLT consists of several parts:
  * Learning: Participants are read a list of 15 unrelated words (List A) in five consecutive trials.
  * Delayed Recall: The participant is asked to recall and repeat back the words from List A. To establish the score for this test, the following elements are considered to calculate the scores:
    * Total learning score: The total number of words correctly recalled in the five trials of List A is added up. Normal scores are 6 words correctly recalled in the first trial and 12 or 13 in the fifth trial. This reflects the ability for learning and short-term memory.
    * Delayed Recall: The number of words recalled from List A after the time interval without practice (20-30 minutes) is noted. This assesses long-term memory. The score can range from 0 to 15 points.
Trail Making Test (TMT) | Up to fourteen days
  It is used to assess executive function and specifically measures timed motor and visual tasks. This test is divided into two parts: Part A (TMT-A), which assesses psychomotor attention and speed and consists of connecting consecutively numbered circles; and Part B (TMT-B), which is based on connecting alternating circles of letters and numbers and measures executive function. A longer time spent completing the test is interpreted as worse performance.
The Digit Symbol Substitution Test (DSST) | Up to fourteen days
  Is a paper-and-pencil cognitive test presented on a single sheet of paper that requires the subject to match symbols to numbers according to a key located at the top of the page. The subject copies the symbol into spaces below a row of numbers. Scoring is based on the number of correct symbols the participant manages to substitute in 90 seconds of time.
Stroop Color and Word Test | Up to fourteen days
  It is used to assess selective attention. This test has a total of 3 slides, each lasting 45 seconds, with a total time of 5 minutes to complete the entire test. In order to read each slide correctly, it must be read from top to bottom and from left to right. The first slide (Stroop Word) is made up of 100 words in which the words "RED", "BLUE" and "GREEN" are repeated, ordered randomly and printed in black ink. This part assesses the number of words read in 45 seconds. After this time, participants must circle the last word they have read. The second slide (Stroop Color) is made up of 100 identical elements "XXXX" in blue, red and green ink. The participant must name the colour of "XXXX" as quickly as possible. Finally, the third slide (Stroop Word-Color) consists of 100 written words that refer to a colour, but are printed in a different colour. Participants must say the color of the ink each word is written in. Higher scores indicate better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Atlántico Medio, Las Palmas de Gran Canaria, Spain